CLINICAL TRIAL: NCT07292103
Title: Effects of Trauma Exposure and Childhood Trauma on Function and Quality of Life in Patients With Temporomandibular Joint Disorders
Brief Title: Trauma Exposure and Childhood Trauma in Temporomandibular Joint Disorders
Status: Completed | Type: Observational
Sponsor: Gulseren Demir Karakilic (Other)
Collaborators: Bozok University (Other); Gaziantep City Hospital (Other)
Responsible Party: Sponsor-Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Other Study IDs: 197/2025
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Disorder; Temporomandibular Joint Dysfunction; Trauma Exposure; Childhood Traumas; Psychological Distress; Quality of Life Impairment
Keywords: Temporomandibular Joint Disorder; Temporomandibular Disorder; Temporomandibular Dysfunction; Mandibular Function Impairment Questionnaire; Hospital Anxiety and Depression Scale; International Trauma Exposure Measure; Childhood Trauma Questionnaire; Short Form-36 Health Survey; Trauma Exposure; Childhood Maltreatment; Adverse Childhood Experiences; Anxiety; Depression; Psychosocial Factors; Quality of Life
MeSH Terms: conditions — Temporomandibular Joint Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Temporomandibular Disorder Group: Adults aged 18 to 65 years with a clinical diagnosis of temporomandibular disorder were included. Participants were cognitively competent, literate, and provided written informed consent. All participants completed structured interviews and standardized questionnaires, including the Mandibular Function Impairment Questionnaire, the Hospital Anxiety and Depression Scale, the International Trauma Exposure Measure, the Childhood Trauma Questionnaire, and the Short Form 36 Health Survey.
- Healthy Control Group: Adults aged 18 to 65 years without a clinical diagnosis of temporomandibular disorder were included. The control group was matched to the patient group according to age and sex. All participants were cognitively competent, literate, and provided written informed consent. Participants in the control group completed the same structured interviews and standardized questionnaires as the patient group, including the Mandibular Function Impairment Questionnaire, the Hospital Anxiety and Depression Scale, the International Trauma Exposure Measure, the Childhood Trauma Questionnaire, and the Short Form 36 Health Survey.

SUMMARY:
Temporomandibular disorder is a multifactorial condition that involves the temporomandibular joint, masticatory muscles, and surrounding structures and is influenced by biological, psychological, and social factors. Parafunctional habits, bruxism, trauma, and occlusal discrepancies have been recognized as important etiological contributors, while psychosocial stressors and early life experiences also play a critical role. Adverse childhood experiences, including neglect and abuse, have been identified as risk factors for long-term psychological vulnerability and physical health problems. Trauma exposure throughout life may further increase the risk of temporomandibular symptoms and negatively affect functional outcomes and quality of life.

The present prospective, cross-sectional case-control study aims to investigate the frequency and impact of childhood trauma and lifetime trauma exposure on functional outcomes and health-related quality of life in patients with temporomandibular disorder. A clinical sample of patients diagnosed with temporomandibular disorder is compared with healthy individuals matched for age and sex. All participants complete standardized questionnaires assessing mandibular function, symptoms of anxiety and depression, cumulative trauma exposure across childhood, adolescence, and adulthood, childhood maltreatment, and health-related quality of life.

By systematically integrating validated measures of both early and later traumatic experiences, this study seeks to provide a comprehensive understanding of the contribution of trauma to the severity and psychosocial burden of temporomandibular disorder. The findings are expected to emphasize the importance of incorporating trauma screening and psychological assessment into the routine evaluation and multidisciplinary management of patients with temporomandibular disorder.

DETAILED DESCRIPTION:
Temporomandibular disorder encompasses a spectrum of neuromuscular and musculoskeletal conditions affecting the temporomandibular joint, masticatory muscles, and related structures. Although its etiology is complex, psychological and social factors have been shown to strongly influence symptom severity and persistence. Previous studies have demonstrated associations between temporomandibular disorder, anxiety, depression, and somatization. Childhood trauma and lifetime traumatic experiences are important determinants of long-term psychological and physical health. However, limited research has investigated the combined influence of adverse childhood experiences and cumulative trauma exposure on functional impairment and quality of life in patients with temporomandibular disorder.

This study was designed to evaluate the prevalence and impact of childhood trauma and lifetime trauma exposure on mandibular function and quality of life in patients with temporomandibular disorder compared with healthy controls.

Study Design

This is a prospective, cross-sectional, observational, case-control study conducted between May 2025 and October 2025. The study protocol was approved by the Human Research Ethics Committee (Approval No: 197/2025). Written and verbal informed consent was obtained from all participants prior to enrollment.

Participants

The patient group consists of adults aged 18 to 65 years with a clinical diagnosis of temporomandibular disorder who are cognitively competent, literate, and willing to participate. The control group consists of healthy individuals without a diagnosis of temporomandibular disorder who are matched with the patient group for age and sex. Control participants are also required to be cognitively competent, literate, and willing to provide informed consent.

Data Collection and Assessments

Data are collected through structured, face-to-face interviews conducted by trained researchers at the otorhinolaryngology outpatient clinic of Gaziantep City Hospital. Participants complete a sociodemographic questionnaire and the following validated assessment instruments:

Mandibular Function Impairment Questionnaire: A seventeen-item self-report measure assessing functional limitations of the mandible, with higher scores indicating greater impairment.

Hospital Anxiety and Depression Scale: A fourteen-item questionnaire assessing symptoms of anxiety and depression through two separate subscales.

International Trauma Exposure Measure: A checklist used to identify exposure to potentially traumatic events across childhood, adolescence, and adulthood. It provides subscale scores for each developmental stage as well as a cumulative lifetime trauma score.

Childhood Trauma Questionnaire: A twenty-eight-item instrument assessing retrospective experiences of childhood maltreatment across five domains, including physical abuse, emotional abuse, sexual abuse, physical neglect, and emotional neglect.

Short Form 36 Health Survey: A thirty-six-item questionnaire evaluating health-related quality of life across eight domains, including physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health.

All instruments are administered in person by the same research team to ensure consistency, reliability, and minimization of measurement bias.

ELIGIBILITY:
Inclusion Criteria

Adults aged 18 to 65 years

Clinically diagnosed with temporomandibular disorder according to standardized clinical evaluation

Cognitively competent and literate individuals capable of completing questionnaires

Voluntary agreement to participate and provision of written informed consent

Exclusion Criteria

History of neurological, psychiatric, or systemic diseases that may affect study participation or data reliability

Cognitive impairment that prevents completion of questionnaires

History of major maxillofacial surgery or trauma not related to temporomandibular disorder

Current substance abuse or alcohol dependence

Refusal or inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included adults aged 18 to 65 years who were recruited from the Otorhinolaryngology outpatient clinic of Gaziantep City Hospital, Türkiye. The patient group consisted of individuals who were clinically diagnosed with temporomandibular disorder, while the control group comprised healthy volunteers without a diagnosis of temporomandibular disorder who were matched to the patient group for age and sex. All participants were cognitively intact, literate, and provided written informed consent prior to participation.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
International Trauma Exposure Measure | At baseline
  The International Trauma Exposure Measure is a standardized checklist designed to evaluate exposure to potentially traumatic events according to the definition of trauma in the International Classification of Diseases, Eleventh Revision. The instrument assesses trauma exposure across three developmental periods: childhood (0-12 years), adolescence (13-18 years), and adulthood (older than 18 years). Subscale scores are calculated separately for each developmental period, and a cumulative lifetime trauma score is obtained by summing all reported events across the lifespan. The Turkish version of the International Trauma Exposure Measure has been validated and demonstrates strong reliability and psychometric properties.
Childhood Trauma Questionnaire | At baseline
  The Childhood Trauma Questionnaire is a 28-item self-report instrument that retrospectively assesses experiences of childhood maltreatment. It consists of five subscales: physical abuse, emotional abuse, sexual abuse, physical neglect, and emotional neglect. Three additional items assess denial or minimization of abuse. Each item is scored on a five-point Likert scale ranging from 1 (never true) to 5 (very often true). Higher subscale and total scores indicate greater severity of childhood trauma. The Turkish adaptation of the Childhood Trauma Questionnaire has been validated and has demonstrated high internal consistency and test-retest reliability.

SECONDARY OUTCOMES:
Mandibular Function Impairment Questionnaire | At baseline
  The Mandibular Function Impairment Questionnaire is a 17-item self-report questionnaire that evaluates perceived limitations in mandibular function. Each item is rated on a five-point Likert scale ranging from 0 (no difficulty) to 4 (very severe difficulty). Total scores range from 0 to 68, with higher scores indicating greater functional impairment. The questionnaire assesses functional limitations during activities such as chewing, speaking, yawning, and other daily tasks. The Turkish adaptation of the Mandibular Function Impairment Questionnaire has been validated and shown to have high reliability and validity.
Hospital Anxiety and Depression Scale | At baseline
  The Hospital Anxiety and Depression Scale is a 14-item questionnaire comprising two subscales: anxiety (7 items) and depression (7 items). Each item is scored from 0 to 3, yielding subscale scores ranging from 0 to 21. Higher scores indicate greater symptom severity. Cut-off values for the depression subscale are defined as follows: 0-7 (normal), 8-10 (mild), 11-14 (moderate), and 15-21 (severe). Similar cut-off values are applied to the anxiety subscale. The Turkish version of the Hospital Anxiety and Depression Scale has been validated and demonstrates good reliability.
Short Form 36 Health Survey | At baseline
  The Short Form 36 Health Survey is a 36-item instrument that assesses health-related quality of life across eight domains: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Each domain is scored on a scale from 0 to 100, with higher scores indicating better perceived health status. The Turkish version of the Short Form 36 Health Survey has been validated and shown to have strong reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (individual participant data) collected during this study, including all de-identified questionnaire and assessment data related to temporomandibular disorder, trauma exposure, childhood experiences, and quality of life, will be made available by the corresponding author upon reasonable request for research purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data and supporting documents will be available after publication of the study results and will remain accessible for five years following publication.
Access Criteria: Researchers who submit a scientifically sound proposal may request access to the de-identified dataset for academic and non-commercial use. Requests should be submitted to the corresponding author via email. Access will be granted following institutional and ethical approval through a secure data-sharing process.
URL: https://hastane.bozok.edu.tr/

REFERENCES:
- [Background] Kocyigit, H., Turkish validity and reliability of short-form 36. Drug Treat, 1999. 12: p. 102-106
- [Background] Şar, V., P.E. ÖZTÜRK, and E. İkikardeş, Çocukluk çağı ruhsal travma ölçeğinin Türkçe uyarlamasının geçerlilik ve güvenilirliği. Turkiye Klinikleri Journal of Medical Sciences, 2012. 32(4): p. 1054-1063.
- [Background] Gündoğmuş, İ., et al., Psychometric properties of the Turkish version of the International Trauma Questionnaire. Journal of Aggression, Maltreatment & Trauma, 2023. 32(12): p. 1847-1865.
- [Background] Hyland P, Karatzias T, Shevlin M, McElroy E, Ben-Ezra M, Cloitre M, Brewin CR. Does requiring trauma exposure affect rates of ICD-11 PTSD and complex PTSD? Implications for DSM-5. Psychol Trauma. 2021 Feb;13(2):133-141. doi: 10.1037/tra0000908. Epub 2020 Sep 10. PMID 32915045
- [Background] Aydemir, Ö., et al., Validity and reliability of Turkish version of hospital anxiety and depression scale. Turk Psikiyatri Derg, 1997. 8(4): p. 280-7.
- [Background] Kılınç, H.E., et al., Further Validity and Reliability of Turkish Version of the Mandibular Functional Impairment Questionnaire in Patients with Temporomandibular Dysfunction. Journal of Basic and Clinical Health Sciences, 2022. 7(1): p. 214-222.